CLINICAL TRIAL: NCT06011187
Title: "Personalized Fluid Administration Using an AFM System for Goal Directed Fluid Therapy on Postoperative Outcome in High-risk Patients Undergoing High-risk Abdominal Surgery: A Multicenter Stepped-wedge, Cluster-randomized Clinical Trial
Brief Title: Assisted Fluid Management (AFM) System and Postoperative Outcome After High-risk Abdominal Surgery
Acronym: PEFLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP220817
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Decision Support System; Outcome
Keywords: hemodynamic; fluid administration; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded and a data monitoring willbe done on data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine care (Active Comparator): During the pre-implementation period, fluid therapy will be done as routine care.
  Mean arterial pressure (MAP) will be maintained between 65-70 mmHg per standard of care
  Interventions: Procedure: Routine care
- Assisted fluid management system (Experimental): In the post-implementation period, fluid bolus administration will be guided by the AFM recommandation.
  MAP will be maintained between 65-70 mmHg per standard of care
  Interventions: Device: AFM

INTERVENTIONS:
Procedure: Routine care — Fluid administration will be given per routine care MAP between 65 - 70 mmHg
  Arms: Routine care
Device: AFM — AFM will recommand fluid bolus administration and MAP will be maintained between 65 and 70 mmHg
  Arms: Assisted fluid management system

SUMMARY:
Goal directed fluid therapy (GDFT) or "Personalized fluid therapy" may benefit high-risk surgical patients but these strategies are infrequently implemented. It has also been shown that without any goal or protocol for fluid resuscitation, large inter- and intra-provider variability exist that have been correlated with poor patient outcomes.

Recently, an "Assisted Fluid Management" (AFM) system has been developed to help ease some of the work associated with GDFT protocol implementation. The AFM system may help increase GDFT protocol adherence while leaving direction and guidance in the hands of the care providers. This artificial intelligence-based system can suggest administration of fluid boluses, analyse the hemodynamic effects of the bolus, and continually re-assess the patient for further fluid requirements.

To date, there are no large outcome study using this AFM system. The primary objective of this trial is thus to evaluate the impact of this AFM system to guide fluid bolus administration on a composite of major postoperative complications in high-risk patients undergoing high-risk abdominal surgery.

DETAILED DESCRIPTION:
Many trials have indicated that goal-directed fluid therapy (GDFT) strategies or more recently "personalized fluid therapy" may benefit high-risk surgical patients but these strategies are infrequently implemented. It has also been shown that without any goal or protocol for fluid resuscitation, large inter- and intra-provider variability exist that have been correlated with poor patient outcomes. Even under ideal study conditions, strict adherence to GDFT protocols is hampered by the workload and concentration required for consistent implementation. Hemodynamic monitors and protocols alone do not enable optimal fluid titration to be provided consistently to all patients - there must also be appropriate and timely interpretation and intervention.

To address this problem of consistency and protocol adherence, a decision support system, "Assisted Fluid Management" (AFM), has been developed to help ease some of the work associated with GDFT protocol implementation. The AFM system (released on the European market in March 2017) may help increase GDFT protocol adherence while leaving direction and guidance in the hands of the care providers. This artificial intelligence-based system can suggest administration of fluid boluses, analyse the hemodynamic effects of the bolus, and continually re-assess the patient for further fluid requirements.

This system was recently implemented in a before-and-after study in a Belgian academic hospital, where the authors reported that the implementation of this AFM software system allowed a better adherence to the GDFT algorithm. However, as this was a pilot study with a small number of patients, the study was not powered to demonstrate a beneficial effect on the incidence of postoperative complications. More recently, a group from the Cleveland Clinic demonstrated that using AFM system resulted in more boluses being effective when compared to the administration of boluses without AFM support.

There are no randomized controlled studies to date comparing this AFM system to standard of care on patient outcome. We therefore aim to conduct a multicenter stepped-wedge, cluster-randomized trial involving patients undergoing high risk abdominal surgery to compare a GDFT strategy guided by the AFM system with usual care.

A stepped wedge, cluster-randomized trial approach was chosen in which clusters will be randomized to commence the intervention at different times following an initial control period in which outcomes will be measured for usual care.

So, each center (cluster) began in the control phase and transitioned to the intervention phase at a randomly assigned time (wedge). The order in which each center will move from control to intervention phase will be randomly allocated by a computer algorithm performed by the study statistician.

We selected cluster randomization rather than randomization of individual patients because the control group could be very different among centers (from GDFT strategy using a flow monitoring to GDFT with a written protocol to no clear strategy (use of an arterial line only without any advanced monitoring). Interestingly, this approach also decreases the Hawthorne effect which has been shown to decrease the incidence rate of the primary outcome in recent randomized trials because clinicians know that their patients are included in a research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient (aged 18 years or older) admitted to the operating room for an elective high-risk abdominal surgery (both open and laparoscopically assisted).
* Patients must fulfill at least one of the following high-risk criteria:
* American Society of Anesthesiologists physical status > 2
* classification exercise tolerance < 4 metabolic equivalents as defined by the guidelines of the American College of Cardiology/ American Heart Association
* renal impairment (serum creatinine ≥1.3mg/dL or >115 mmol/l or estimated glomerular filtration rate < 90 mL/min/1.73 m2 within the last 6 months) or renal replacement therapy
* coronary artery disease (any stage)
* chronic heart failure (New York Heart Association Functional Classifcation ≥ II)
* valvular heart disease (moderate or severe);
* history of stroke
* peripheral arterial occlusive disease (any stage)
* chronic obstructive pulmonary disease (any stage) or pulmonary fibrosis (any stage)
* diabetes mellitus requiring oral hypoglycemic agent or insulin; immunodeficiency due to a disease (e.g., HIV, leukemia, multiple myeloma, solid organ cancer) or therapy (e.g., immunosuppressants, chemotherapy, radiation, steroids)
* liver cirrhosis (any Child-Pugh class)

  -- body mass index ≥30 kg/m2
* current smoking or 15 pack-year history of smoking
* All participants must receive clear study information and give signed informed consent

Exclusion Criteria:

* Patients with preoperative cardiac arrhythmias (atrial fibrillation) as the monitoring devices are not accurate under cardiac arrhythmias.
* No affiliation with the French health care system
* Patients participating in another randomized controlled trial with the same clinical endpoint, or interventions possibly compromising the primary outcome.
* Pregnant patients
* Patient on AME (state medical aid) (unless exemption from affiliation)
* Patients guardianship/legal protection/curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint ("any event versus none") of major postoperative complications within 30 days after surgery | Postoperative day 30
  It includes : acute myocardial injury, including myocardial infarction, acute kidney injury, severe infectious complications (including deep surgical site infection, pneumonia, sepsis, peritonitis), anastomotic leakage, pulmonary embolism or venous thrombosis, pulmonary edema, acute respiratory distress syndrome, de novo arrhythmia, stroke, reoperation for any cause, non-fatal cardiac arrest, and mortality within 30 days after surgery

SECONDARY OUTCOMES:
Incidence of each of the individual components of the composite primary outcome within 30 days after surgery | Postoperative day 30
Incidence of the composite primary outcome within 7 days after surgery | Postoperative day 7
Incidence of a composite of postoperative infection rate within 30-day of surgery. | Postoperative day 30
  This is defined as one or more of the following infections: surgical site infection, organ space surgical-site infection, urinary tract infection, laboratory-confirmed blood stream infection or infection, source uncertain (this is defined as an infection which could be more than one of the above but it is unclear which)
Clavien-dindo classification score | Postoperative day 30
Comprehensive complication index (CCI) | Postoperative day 30
Length of stay in the hospital | Postoperative day 30
Incidence of unplanned hospital re-admission within 30 days after surgery | Postoperative day 30
Mortality rate at 90 days after surgery. | Postoperative day 90

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDRE JOOSTEN, MD PhD, Study Director — PAUL BROUSSE HOSPITAL
Locations (17):
- United States (2):
  - University of California IRVINE, Irvine, California
  - University of California Los Angeles (UCLA), Los Angeles, California
- UZ Brussels, Brussels, Brussels Capital, Belgium
- CHUM Montreal, Montreal, Montreal, Canada
- France (12):
  - Chu Dijon, Dijon, Dijon
  - ALEXANDRE JOOSTEN, MD PhD, Le Kremlin-Bicêtre, France
  - Chu Grenoble Alpes, Grenoble, Grenoble
  - Centre chirurgical Marie Lannelongue, Le Plessis-Robinson, Haut de Seine
  - BICETRE, Le Kremlin-Bicêtre, Paris
  - BEAUJON, Paris, Paris
  - HEGP, Paris, PARIS
  - Insititut Mutualiste Montsouris, Paris, Paris
  - La Pitie Salpetriere, Paris, PARIS
  - Chu Toulouse, Toulouse, Toulouse
  - Chu Lille, Lille
  - Centre hospitalier universitaire de NANCY, Nancy
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coeckelenbergh S, Delaporte A, Rousseleau D, De Montblanc J, Roullet S, Ramadan J, Cholley B, Sitbon A, Weiss E, Kassab MC, Diop S, Manzi E, Pustetto M, Porta Bonette G, Guinot PG, Guerci P, Vanhonacker D, Carrier FM, Alexander B, Rinehart J, Boldt D, Grogan T, Cannesson M, Duranteau J, Grimaldi L, Pereira B, Joosten A. Investigating the effectiveness of an intraoperative decision support guided fluid therapy intervention on postoperative outcome of high-risk patients undergoing high-risk abdominal surgery: protocol for an international multicentre stepped-wedge cluster-randomised implementation trial. BJA Open. 2025 Jun 5;14:100421. doi: 10.1016/j.bjao.2025.100421. eCollection 2025 Jun. PMID 40529718